CLINICAL TRIAL: NCT05875597
Title: Detection of Clinical-functional Changes Following Exercise Therapy and Education in Institutionalised and Community-dwelling Older Adults Diagnosed With Sarcopenia
Brief Title: Detection of Clinical-functional Changes Following Exercise Therapy and Neuroscience Education in Institutionalised and Community-dwelling Older Adults Diagnosed With Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Luis Espejo Antunez, Ph.D. Physical Therapy, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEAntunez
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-02

CONDITIONS: Resistance Training; Aged; Nursing Homes; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group Exercise (Experimental): Participants will be required to undertake a strength oriented physical therapy exercise programme.
  Interventions: Other: Physical therapy exercise programme
- Control Group (No Intervention): Participants will not engage in a strength oriented therapeutic physical exercise programme.

INTERVENTIONS:
Other: Physical therapy exercise programme — Carrying out a programme of therapeutic physical exercise for 12 weeks, twice a week for 45 minutes.
  Arms: Experimental Group Exercise

SUMMARY:
Nowadays, ageing is an important aspect to consider from a social, healthcare and economic perspective. For this reason, it is necessary to focus on all the elements which can help staying healthy and active in old age. Physical activity and exercise are one of these, and more specifically resistance training.

DETAILED DESCRIPTION:
Recently, it is been evidenced that physical activity and exercise are an important coping strategy to get what is called "active ageing". However, it is still under discussion some key aspect, like the training type or the optimal dose, among others. There is a modality of resistance training which it has not been sufficiently studied in old age population: the high intensity interval training. It has been demonstrated in other population (like cardiovascular patients or cancer survivor patients) that this modality of training can improve a lots their physical condition. Furthermore, it produces a higher adhesion to the training program, because it does not require so long time like another type of training. For this reason, the aim of this investigation is to assess how implement this modality of training on elderly people with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 55 years or older.
* Living in an institutionalised setting or community-dwelling older adults living in the province of Badajoz or Cáceres.
* Voluntarily participating in the study.
* Who had a diagnosis of sarcopenia/fragility in the last year.
* Submit a prescription from the centre's medical practitioner to participate in the study as physiotherapy intervention would be appropriate and potentially beneficial.

Exclusion Criteria:

* Patients with cognitive impairment (score ≥24 in the validated Spanish version for general older adults of the Mini-Mental Status Examination).
* Unable to tolerate moderate physical activity due to cardiovascular or respiratory disease.
* With balance disorders other than those caused by ageing such as dizziness or vestibular disorders requiring the ingestion of medication with a potential effect on balance, as well as balance disorders secondary to the ingestion of any medication or other medical causes.
* At high risk of falling (≥ 51 points on the MORSE scale).
* At high risk of falling (≥ 51 points on the MORSE scale).
* At high risk of falling (≥ 51 points on the MORSE scale).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes in handgrip strength | 12 weeks
  Hand-held dynamometer JAMAR
Changes in muscle mass | 12 weeks
  electrical bioimpedance
Changes in physical performance | 12 weeks
  SPPB test battery
Changes in Funcional Mobility | 12 weeks
  Measured by the Timed Up and Go test (TUG)

SECONDARY OUTCOMES:
Changes in Risk of falling | 12 weeks
  The Downton, Tinetti fall risk index was used to assess the risk of falling.
Changes in Health-Related Quality of Life | 12 weeks
  Will be measured through the SF-12 health questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo Antúnez, Study Director — Universidad de Extremadura
Locations (1):
- Rosalba Nursing Home, Mérida, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benavent-Caballer V, Sendin-Magdalena A, Lison JF, Rosado-Calatayud P, Amer-Cuenca JJ, Salvador-Coloma P, Segura-Orti E. Physical factors underlying the Timed "Up and Go" test in older adults. Geriatr Nurs. 2016 Mar-Apr;37(2):122-7. doi: 10.1016/j.gerinurse.2015.11.002. Epub 2015 Dec 17. PMID 26707544
- [Background] Pagotto V, Nakatani AY, Silveira EA. [Factors associated with poor self-rated health in elderly users of the Brazilian Unified National Health System]. Cad Saude Publica. 2011 Aug;27(8):1593-602. doi: 10.1590/s0102-311x2011000800014. Portuguese. PMID 21877007
- [Background] Fielding RA, Vellas B, Evans WJ, Bhasin S, Morley JE, Newman AB, Abellan van Kan G, Andrieu S, Bauer J, Breuille D, Cederholm T, Chandler J, De Meynard C, Donini L, Harris T, Kannt A, Keime Guibert F, Onder G, Papanicolaou D, Rolland Y, Rooks D, Sieber C, Souhami E, Verlaan S, Zamboni M. Sarcopenia: an undiagnosed condition in older adults. Current consensus definition: prevalence, etiology, and consequences. International working group on sarcopenia. J Am Med Dir Assoc. 2011 May;12(4):249-56. doi: 10.1016/j.jamda.2011.01.003. Epub 2011 Mar 4. PMID 21527165
- [Background] Brocca L, McPhee JS, Longa E, Canepari M, Seynnes O, De Vito G, Pellegrino MA, Narici M, Bottinelli R. Structure and function of human muscle fibres and muscle proteome in physically active older men. J Physiol. 2017 Jul 15;595(14):4823-4844. doi: 10.1113/JP274148. Epub 2017 Jun 5. PMID 28452077
- [Background] Servais S, Letexier D, Favier R, Duchamp C, Desplanches D. Prevention of unloading-induced atrophy by vitamin E supplementation: links between oxidative stress and soleus muscle proteolysis? Free Radic Biol Med. 2007 Mar 1;42(5):627-35. doi: 10.1016/j.freeradbiomed.2006.12.001. Epub 2006 Dec 15. PMID 17291986
- [Background] Narici MV, Maffulli N. Sarcopenia: characteristics, mechanisms and functional significance. Br Med Bull. 2010;95:139-59. doi: 10.1093/bmb/ldq008. Epub 2010 Mar 2. PMID 20200012
- [Background] Dietzel R, Felsenberg D, Armbrecht G. Mechanography performance tests and their association with sarcopenia, falls and impairment in the activities of daily living - a pilot cross-sectional study in 293 older adults. J Musculoskelet Neuronal Interact. 2015 Sep;15(3):249-56. PMID 26350943
- [Background] Cederholm T, Cruz-Jentoft AJ, Maggi S. Sarcopenia and fragility fractures. Eur J Phys Rehabil Med. 2013 Feb;49(1):111-7. PMID 23575205

DOCUMENTS (1):
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT05875597/ICF_000.pdf